CLINICAL TRIAL: NCT01875341
Title: Resistant Hypertension in Patient With Diabetic Nephropathy: Role of Sleep Apnea and Associated Sympathetic Hyperactivity.
Brief Title: Role of Sleep Apnea and Sympathetic Activity in Resistant Hypertensive Patients.
Acronym: SAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Marcel Ruzicka, Dr. Marcel Ruzicka, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005972-01H
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes; Diabetic Nephropathy; Hypertension; Sleep Apnea
Keywords: type 2 diabetes; diabetic nephropathy; hypertension; sleep apnea; sympathetic hyperactivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Hypertension; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment with NCPAP (Active Comparator): This group will receive treatment with NCPAP, Nasal Continuous Positive Airway Pressure for 6 weeks. Nasal Continuous Positive Airway Pressures will be increased until apneas & hypopneas are prevented during all sleep stages.
  Interventions: Device: NCPAP; Nasal continuous positive airway pressure.; Device: NCPAP Nasal Continuous Positive Airway Pressure-sub-therapeutic treatment group
- Sub- active treatment with NCPAP (Sham Comparator): This group will receive treatment with Nasal Continuous Positive Airway Pressure at sub-therapeutic levels for 6 weeks. Patients will be taught how to use NCPAP in the sleep lab. Pressures will be left unchanged at the lowest possible value for the NCPAP device. After completion of treatment patients will be provided usual NCPAP therapy.
  Interventions: Device: NCPAP; Nasal continuous positive airway pressure.; Device: NCPAP Nasal Continuous Positive Airway Pressure-sub-therapeutic treatment group

INTERVENTIONS:
Device: NCPAP; Nasal continuous positive airway pressure. — Patients will be randomized to receive either therapeutic or sub-therapeutic NCPAP; Nasal continuous positive airway pressure treatment. In patients randomized to therapeutic NCPAP, treatment pressures will be increased until apneas and hypopneas are prevented during all sleep stages. In the sub-therapeutic treatment group, pressure will be left unchanged at the lowest possible value for the NCPAP device. Pressure settings for NCPAP therapy will be determined by Dr. J. Leech, collaborator and specialist in sleep disorders. Treatment will be continued for a total of 6 weeks.
Device: NCPAP Nasal Continuous Positive Airway Pressure-sub-therapeutic treatment group — In the sub-therapeutic treatment group, pressure will be left unchanged at the lowest possible value for the NCPAP device. Pressure settings for NCPAP therapy will be determined by Dr. J. Leech, collaborator and specialist in sleep disorders. Treatment will be continued for a total of 6 weeks.

SUMMARY:
Hypertension is highly prevalent in type 2 diabetic patients (NIDDM) with nephropathy, and is the single most important determinant of the rate of renal function loss. In many of these patients, hypertension is resistant to therapy. Although increased sympathetic activity is also highly prevalent in NIDDM patients with nephropathy and chronic renal insufficiency, little attention has been paid to sleep apnea as the cause of both resistant hypertension and sympathetic hyperactivity in this population. Since the prevalence of sleep apnea is increased in patients with either NIDDM, or resistant hypertension, or chronic renal insufficiency, it is almost certain that sleep apnea has a high prevalence in patients in whom all three states co-exist, i.e. NIDDM patients with nephropathy and hypertension resistant to therapy. As a consequence of undetected and untreated sleep apnea, resistant hypertension, nocturnal hypertension, and sympathetic hyperactivity likely contribute to accelerated loss of renal function and increased cardiovascular morbidity and mortality in these patients.

Hypothesis: A. Sleep apnea is highly prevalent in type 2 diabetic patients with diabetic nephropathy and hypertension resistant to therapy. Treatment with nasal continuous positive airway pressure (NCPAP) will result in a decrease in blood pressure and restore normal diurnal blood pressure pattern.

B. Sleep apnea-caused hypertension is mediated by sympathetic hyperactivity and increased activity of the renin-angiotensin-aldosterone system (RAAS) in type 2 diabetic patients with nephropathy. A decrease in sympathetic hyperactivity in response to NCPAP therapy will result in a decrease in plasma renin activity and plasma aldosterone concomitant with decreases in blood pressure.

Randomized, double blind, parallel comparative (two groups) one center trial.

Therapeutic treatment with nasal continuous positive airway pressure (NCPAP) Sub-therapeutic treatment with nasal continuous positive airway pressure

DETAILED DESCRIPTION:
The study will be double blind and consist of two parallel groups. Patients with type 2 diabetes with a creatinine clearance above 20 ml/min and with microalbuminuria or proteinuria who have both resistant hypertension and sleep apnea will be studied. Creatinine clearance and proteinuria will be assessed from a 24 hour urine collection not older than 6 months. Microalbuminuria will be assessed from at least 2 out of 3 positive random urine samples with the last one not older than 6 months. Blood pressure will be considered as resistive to treatment if the patient is on 3 or more antihypertensive medications with blood pressure readings of greater than 140/90 mmHg on the last 2 out of 3 office visits. Sleep apnea syndrome will be defined by the presence of at least 5 apneic or hypopneic episodes per hour during an overnight sleep study.

Screening will be done in the following manner: Patients seen in the Hypertension Unit at the University of Ottawa Heart Institute, General Nephrology Clinic and Progressive Renal Insufficiency Clinic at the Ottawa Hospital, will be screened by the study coordinator. For the patients who meet the study criteria, the attending physician is asked for permission to contact each patient. If patients agree to participate, they will undergo a sleep study. Screening of patients and subsequent sleep studies will continue until 54 consecutive patients with moderate to severe sleep apnea (15 apneic or hypopneic episodes per hr) are found and enrolled into the study. The prevalence of sleep apnea in the specialty clinic population will be calculated as the number of patients with sleep apnea diagnosed based on a sleep study divided by the total number of clinic patients screened who underwent a sleep study.

After the baseline visit and completion of all preliminary procedures, specific studies for microneurography, plasma renin and aldosterone will be performed. Consequently, a 24 hour blood pressure monitor and a 24 hour urine collection for creatinine clearance, microalbuminuria and proteinuria will be done. Once all the testing has been completed, the patient will be randomized to therapeutic or sub-therapeutic treatment with nasal continuous positive airway pressure for 6 weeks. After 6 weeks of treatment the specific studies, 24 hour blood pressure monitoring and 24 hour urine collection will be repeated.

ELIGIBILITY:
Inclusion Criteria:.

1. Males and females 18 years or older
2. On 3 or more antihypertensive medications with resistant hypertension of >140/90 mmHg (resting) despite treatment
3. Diagnosis of sleep apnea (15 apneic/hypopneic episodes per hour and a score of 10 on Epworth sleepiness scale).
4. Creatinine clearance > 20 ml/min with microalbuminuria or proteinuria, (results within past 6 months)

Exclusion Criteria:

1. Acute coronary syndrome within 6 months
2. Patients with clinically documented congestive heart failure
3. Patients with relevant cardiac arrhythmias (second and third-degree heart block or premature ventricular complexes in Lown classes IV or V)
4. Pregnant or lactating women
5. Patients with leg injury involving nerve damage
6. Patients with symptomatic peripheral neuropathy
7. Patients with predominant central sleep apnea
8. Patients mentally unable to give informed consent
9. Professional drivers
10. Patients with a resting blood pressure >180/110 mmHg
11. Patients taking clonidine
12. Patients with sleep apnea causing daily drowsiness
13. Patients with severe hyperkalemia (>5.5 mmol/L) or hypokalemia (<3.3 mmol/L)
14. Patients with a BMI of >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Primary end-point: change in daytime and night-time mean systolic blood pressure | baseline and 6 weeks post intervention
  Blood pressures will be assessed by 24 hour ambulatory blood pressure monitoring (ABPM) from baseline to after 6 weeks of therapy in the two treatment groups

SECONDARY OUTCOMES:
changes in daytime and night-time mean diastolic blood pressure | baseline and post 6 weeks of therapy
  Blood pressures will be assessed by 24 hour blood pressure monitoring
muscle sympathetic nerve activity -microneurography | Baseline and 6 weeks post intervention
  microneurography,will assess sympathetic hyperactivity measuring Muscle sympathetic-nerve activity from the peroneal nerve. A tungsten micro electrode will be inserted into the peroneal nerve. A reference electrode will be placed subcutaneously 1 to 2 cm from the recording electrode. The sympathetic activity will be amplified, filtered, integrated and displayed on a computer monitor. In addition, the signal will be digitized and recorded on a computer with a sampling rate of 2,000 Hz. All recordings will be done in a similar manner after at least 20 minutes of rest and will be combined with continuous blood pressure and heart rate measurements.
  Muscle sympathetic-nerve activity will be expressed as the number of bursts per minute and as the number of bursts per 100 heart beats, to correct for differences in heart rate.
plasma renin and aldosterone | baseline to after 6 weeks
  serum renin and aldosterone levels will be drawn after 30 minutes of rest . All samples will be collected in the appropriate tubes, shielded from the light and immediately placed on ice. Samples will be processed and stored at -80°C for analysis at a later date.
  Plasma renin activity will be assessed by radioimmunoassay (RIA). Plasma aldosterone will be assessed by RIA after separation by High-performance liquid chromatography (HPLC)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, Dr., Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada